CLINICAL TRIAL: NCT03370315
Title: Effects of a Dance and Walking Program on Gait and Quality of Life in People With Parkinson's Disease
Brief Title: Effects of a Dance and Walking Program for People With Parkinson's Disease
Acronym: DANCEPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Aline Nogueira Haas, Principal Investigator, Federal University of Rio Grande do Sul
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DANPD017
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Parkinson Disease
Keywords: Parkinsonian Disorders; Dance Therapy; Rehabilitation; Kinematics; Locomotion; Quality of Life
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dance Group (Experimental): This group will be undergo dance classes two times a week, for 12 weeks. 24 sessions.
  Intervention administered: Dance classes inspired by the rhythm of Forró and Samba.
  Interventions: Other: Dance Program
- Walking Group (Experimental): This group will be undergo walking training two times a week, for 12 weeks. 24 sessions.
  Intervention administered: Walking program with 3 different moments.
  Interventions: Other: Walking Program

INTERVENTIONS:
Other: Dance Program — The dance program consists of dance classes inspired by the rhythm of Forró and Samba. The sessions are divided into four stages: 1) stretching and sensitization of the body, with the support of chairs; 2) balance and rhythm exercises, with the support of the bar; 3) dance inspired by the genres worked - Forró and Samba; 4) Fun activities that stimulate socialization or with visual clues, working displacements, motor coordination, rhythm, improvisation and creativity. 24 sessions, twice a week, which session take 60 min.
  Arms: Dance Group
Other: Walking Program — The walking program consists of 3 moments: 1) a brief warm-up of free walking for 3 minutes in the comfortable velocity; 2) then walking according to the training cycle, the intensity will be between 60 and 80% of the reserve heart rate; 3) a relaxation. 24 sessions, twice a week, which session take 60 min.
  Arms: Walking Group

SUMMARY:
Parkinson's disease (PD), characterized as progressive and neurodegenerative, is one of the most frequent neurological diseases of the present time. Patients with PD present motor impairment, such as muscle stiffness, rest tremor, slow movements, postural instability, and gait and balance alterations; And non-motor factors, such as cognitive and neuropsychiatric disorders, depressive symptoms, and a consequent decrease in quality of life (QL). Dance can be an important tool for the complementary treatment of these patients, when added to traditional drug therapies and physiotherapies. Thus, the present study aims to verify the effects of a program of dance and walking in gait and QL of 38 adults with PD, divided in two groups, and to compare the aspects of functionality, dynamic stability, kinematics and QL. The data collection instruments will be a personal data sheet of the patients, the Hoehn and Yahr Scale (H&Y), the Rehabilitation Index (RI), the motor part of the Unified PD Rating Scale (UPDRS III), the Timed Up ang Go test (TUG), the kinematic analysis of walking and the Parkinson's Disease Questionnaire (PDQ-39). Statistical Package for Social Sciences (SPSS) software version 20.0 will be used to analyze the data, using the Wilcoxon test for non-parametric data and the paired t-test for parametric data, in order to compare pre and post intervention data. The significance level adopted for both tests will be p <0.05. It is expected that a program of 24 sessions of dance classes will be as or more effective than a program of 24 walking sessions for the gait quality and QL for the participants of the study.

ELIGIBILITY:
Inclusion Criteria:

* Both sex;
* Equal to or more than 50 years old;
* Parkinson Disease in regular medical treatment and follow-up;
* Illness diagnosis equal to or more than one year;
* H&Y scale between one and three;
* Able to walk independently or with a walking stick.

Exclusion Criteria:

* More than six absences in dance class or in the walking training (25%);
* Start a new activity parallel to the project;
* Risk factors: Recent surgeries, Deep brain stimulation surgery (DBS), Other associated neurological diseases or other chronic diseases.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
The change in functional mobility | Before and after 12 weeks after the intervention
  The functional mobility will be assessed using the Timed Up and Go Test. This first outcome will be evaluated before and after 12 weeks of Dance Classes and Walking Training in both groups.

SECONDARY OUTCOMES:
The change in the gait specific parameters | Before and after 12 weeks after the intervention
  The gait specific parameters will be assessed using the BTS SMART DX 7000. This secondary outcome will be evaluated before and after 12 weeks of Dance Classes and Walking Training in both groups.
The change in Quality of Life | Before and after 12 weeks after the intervention
  Quality of Life will be assessed using Parkinsons' Disease Questionnaire (PDQ-39). The Quality of Life questionnaire will be evaluated before and after 12 weeks of Dance Classes and Walking Training in both groups. Parkinson's Disease Questionnaire (PDQ39) measures patients' quality of life through 39 questions. The instrument is divided into eight dimensions: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication and bodily discomfort. In total, patients answer 39 questions that should be noted among five response options: "never," "rarely," "sometimes," "often" or "always."
The change in motor symptoms | Before and after 12 weeks after the intervention
  Motor symptoms will be assessed using Unified Parkinsons' Disease Rating Scale (UPDRS). The motor symptoms will be evaluated before and after 12 weeks of Dance Classes and Walking Training in both groups. We will use the Part III of the Unified Parkinson's Disease Rating Scale (UPDRS III), which measures the motor symptoms of the disease. Part III of the UPDRS is composed of 14 items, covering questions 18 to 31 of the scale. Each item has 5 response options that add up to 0 to 4 points, how bigger is the total score on the scale; greater is the patient's motor impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Aline N. Haas, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hackney ME, Kantorovich S, Levin R, Earhart GM. Effects of tango on functional mobility in Parkinson's disease: a preliminary study. J Neurol Phys Ther. 2007 Dec;31(4):173-9. doi: 10.1097/NPT.0b013e31815ce78b. PMID 18172414
- [Result] Cavagna GA, Franzetti P, Heglund NC, Willems P. The determinants of the step frequency in running, trotting and hopping in man and other vertebrates. J Physiol. 1988 May;399:81-92. doi: 10.1113/jphysiol.1988.sp017069. PMID 3404473
- [Result] Shanahan J, Morris ME, Bhriain ON, Saunders J, Clifford AM. Dance for people with Parkinson disease: what is the evidence telling us? Arch Phys Med Rehabil. 2015 Jan;96(1):141-53. doi: 10.1016/j.apmr.2014.08.017. Epub 2014 Sep 16. PMID 25223491
- [Derived] Dos Santos Delabary M, Monteiro EP, Donida RG, Wolffenbuttel M, Peyre-Tartaruga LA, Haas AN. Can Samba and Forro Brazilian rhythmic dance be more effective than walking in improving functional mobility and spatiotemporal gait parameters in patients with Parkinson's disease? BMC Neurol. 2020 Aug 18;20(1):305. doi: 10.1186/s12883-020-01878-y. PMID 32811464